CLINICAL TRIAL: NCT03535324
Title: Opportunities for Antibiotic Optimisation and Outcomes Improvement in Patients With Negative Blood Culture (The NO-BACT Project)
Brief Title: Opportunities for Antibiotic Optimisation and Outcomes Improvement in Patients With Negative Blood Culture (NO-BACT)
Acronym: NO-BACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NO-BACT (FIS-ANT-2018-01)
Record Dates: First submitted 2018-05-08; First posted 2018-05-24 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Antibiotic Resistant Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROA for optimization (Experimental): Development of a Program for optimizing the use of antibiotics (PROA) in Spanish (Antimicrobial Stewardship Program, ASP, in English), based on Reinforcement, Guidance and Support Programs, to prescribing physicians for the optimization of antimicrobial use based on a non-tax counseling program and evidence-based recommendations. The intervention will be carried out at the cluster level (group of patients belonging to a specific hospital service that meet the inclusion criteria). The intervention will consist in carrying out the audit with recommendation on days 3 and 5-7 after the extraction of negative blood cultures to assess the possibilities of de-escalation, sequential oral therapy and end of early treatment based on the available evidence.
  Interventions: Behavioral: PROA for optimization
- Control (Other): There will be no intervention.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: PROA for optimization — The development of a ASP based on Reinforcement, Guidance and Support Programs, to prescribing physicians for the optimization of antimicrobial use based on a non-tax counseling program and evidence-based recommendations.
  Arms: PROA for optimization
Other: Control — There will be no intervention
  Arms: Control

SUMMARY:
Patients with negative blood cultures represent 85-90 % from all patients with a blood culture taken during hospital admissions. This population usually includes an heterogeneous group of patients that are admitted because of an infectious diseases or febrile syndrome in which performing a blood culture is required. There is scarce evidence about the clinical characteristics and the antibiotic treatment given to these patients. This project will be developped in two phases with an specific target in each one:

* Phase I (a cohort study of patient with blood cultured taken): the investigators aim to analyse the clinical and therapeutics characteristics, outcomes and antimicrobial stewardship oppotunities in a population of patients with negative blood culture. The investigators aim to compare the outcomes and antimicrobial stewardship opportunities with those in patients with positive blood culture.
* Phase II: The investigators will develop a cluster randomised control trial to evaluate the implementation of a targeted antimicrobial stewardship intervention in patients with negative blood culture (based on 3rd and 5th day audits). The effect of the intervention on the quality of antimicrobial use (duration and de-escalation), long of stay and mortality will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals in charge of patients with negative hemoculture and active antibiotherapy within 48 hours of extraction; and that belong to a clinical unit that has been assigned to the intervention arm.

Exclusion Criteria:

* Health professionals in charge of patients who, even if they meet the criteria described above, will not be considered to have a foreseeable death within <72hrs from the hemoculture extraction or a positive hemoculture in the seven days prior to the extraction of the negative hemoculture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Days of treatment (DDT) | It will be variable because each individual can have a different treatment days that will vary based on our previous experience between 2 and 28 days . They will be measured only once for each case included.
  Days of treatment per negative hemoculture episode evaluated

SECONDARY OUTCOMES:
Defined Daily Doses (DDDS) | Weekly from date of randomization up to 28 days
  Defined Daily Doses of antibiotic used in each episode
30-day mortality | From 4 to 30 days since only those patients with active antibiotherapy are included at 48 hours and with no death forecast before 48-72 hours after inclusion
  Mortality at 30 days after the extraction of the blood culture.
Re-hospitalization in the next 90 days | From 4 to 90 days
  Re-hospitalization in the next 90 days after the extraction of the blood culture.
Superinfection by multiresistant microorganisms | In the first three months after the negative blood culture
  Rate of reinfection by MDR (multidrug-resistant) bacteria (according to Magiorakos AP et al criteria - International standard definitions for acquired resistance, Clin Microbiol Infect, 2011) among the intervention group patients comparing to rate in the control group patients
Clostridium difficile diarrhea | In the first three months after the negative blood culture
  Rate of patients presenting confirmed Clostridium difficile (CD) diarrhea among the intervention group patients comparing to rate of CD diarrhea about control group patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Retamar Gentil, MD/PhD, Study Director — Virgen Macarena Hospital
Locations (3):
- Spain (3):
  - Puerta del Mar Hospital, Cadiz
  - Virgen Macarena Hospital, Seville
  - Lozano Blesa Hospital, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Jorge S, Palacios-Baena ZR, Rosso-Fernandez CM, Giron-Ortega JA, Rodriguez-Bano J, Retamar P. Opportunities for antibiotic optimisation and outcome improvement in patients with negative blood cultures: study protocol for a cluster-randomised crossover trial, the NO-BACT study. BMJ Open. 2019 Dec 18;9(12):e030062. doi: 10.1136/bmjopen-2019-030062. PMID 31857298